CLINICAL TRIAL: NCT02548858
Title: Perineorrhaphy Outcomes Related to Body Imagery (POETRY)
Brief Title: Perineorrhaphy Outcomes Related to Body Imagery
Acronym: POETRY
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of New Mexico (Other)
Responsible Party: Principal Investigator, Cara Ninivaggio, Urogynecology Fellow, University of New Mexico, University of New Mexico
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 15-108
Record Dates: First submitted 2015-09-08; First posted 2015-09-14 (Estimated); Last update posted 2019-03-04 (Actual); Status verified 2019-03

CONDITIONS: Pelvic Organ Prolapse
Keywords: Perineorrhaphy; Pelvic organ prolapse; Vaginal or abdominal reconstruction; Body image
MeSH Terms: conditions — Pelvic Organ Prolapse

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Perineorrhaphy (Active Comparator): Patients who are randomized to receive a perineorrhaphy as part of their vaginal or abdominal reconstructive procedure
  Interventions: Procedure: Perineorrhaphy
- No Perineorrhaphy (Active Comparator): Patients who are randomized not to receive a perineorrhaphy as part of their vaginal or abdominal reconstructive procedure
  Interventions: Procedure: No Perineorrhaphy

INTERVENTIONS:
Procedure: Perineorrhaphy — Those patients who are randomized to undergo a perineorrhaphy as part of their vaginal or abdominal reconstructive procedure for pelvic organ prolapse.
  Arms: Perineorrhaphy
Procedure: No Perineorrhaphy — Those patients who are randomized not to undergo a perineorrhaphy as part of their vaginal or abdominal reconstructive procedure for pelvic organ prolapse.
  Arms: No Perineorrhaphy

SUMMARY:
The purpose of this study is to determine whether performing a perineorrhaphy during a reconstructive surgery indicated for pelvic organ prolapse (POP) affects a patient's body image.

DETAILED DESCRIPTION:
The objective of this study is to assess the body image of women before and after pelvic reconstructive surgery with and without perineorrhaphy to examine if a perineorrhaphy impacts postoperative body image by conducting a single-blind, randomized controlled clinical trial. The central hypothesis is that patients' body image will not be affected by whether or not a perineorrhaphy is performed.

The target population are those patients with POP who are planning an apical prolapse repair. All participants will give written consent prior to their surgery. After enrollment, women will fill out baseline surveys, including the Body Image in Pelvic Organ Prolapse (BIPOP), the Pelvic organ prolapse/Incontinence Sexual Questionnaire, IUGA-revised) (PISQ-IR), the Pelvic Floor Distress Inventory (PFDI-20), and a Pain Visual Analog Scale (VAS) to assess baseline pain. Additionally, participants will undergo a Pelvic Organ Prolapse Quantification (POP-Q) examination with the addition of measurements of genital hiatus (GH) and perineal body (PB) lengths without strain. The other measurements involved in the POP-Q entail assigning numerical values to descent of different parts of the vagina. Pelvic floor muscle strength will be measured using a Peritron™ perineometer and Kegel strength (contraction of the pelvic floor muscles) using the Oxford grading scale.

On the day of the patient's surgery, the surgeon will call a research coordinator who will open the next envelope in the sequence randomizing the patient to perinorrhaphy or to no perineorrhaphy. Randomization assignment will be generated by a computer-based randomization table and assigned by a research coordinator not otherwise involved in the study. Women will not be informed to what arm of the study they were randomized, and postoperative assessments will be made by individuals not involved with the patient's surgery.

At prescribed time points post-operatively, the patients will be assessed by POP-Q, genital hiatus and perineal body measurements performed with and without strain, the pain VAS, the BIPOP, The PISQ-IR, the PFDI-20, and pelvic floor muscle strength via the Oxford scale and measurement by the Peritron™ perineometer.

The investigators' aims for this study are:

Aim #1: To determine if a patient's body image, by using the Body Image in Pelvic Organ Prolapse (BIPOP) questionnaire, is affected by concomitant performance of a perineorrhaphy at the time of pelvic organ prolapse surgery. Hypothesis: There will be no difference in body image scores between those with and without concomitant perineorrhaphy.

Aim #2: To determine if Pelvic Organ Prolapse Quantification (POP-Q) measurements are affected by a perineorrhaphy. Hypothesis: After a perineorrhaphy, the genital hiatus (GH) will be smaller, the total vaginal length (TVL) will be longer, the perineal body (PB) will be longer, and all others will be unaffected when compared to those in whom perineorrhaphy is not performed.

Aim #3: To determine if the strength of pelvic floor muscles is improved after corrective pelvic organ prolapse surgery with a perineorrhaphy compared with those patients who did not have a perineorrhaphy, as measured by the Peritron™, a perineometer device that measures pelvic floor muscle contraction strength. Hypothesis: Pelvic floor muscle strength will be unaffected by the performance of a perineorrhaphy.

Aim #4: To assess if those having a perineorrhaphy have higher postoperative pain both in the short term and long term by using a visual analog scale (VAS) both in the immediate and 6 week postoperative period. Hypothesis: Those with perineorrhaphies will report more pain on a VAS both immediately and 6 weeks post-surgery.

Aim #5: To describe if there are differences in sexual function after corrective pelvic organ prolapse with a perineorrhaphy compared to those who did not undergo a perineorrhaphy. Hypothesis: Sexual function will be improved after POP surgery repair but will be unaffected by the performance of a perineorrhaphy.

ELIGIBILITY:
Inclusion Criteria:

* Subjects ≥ 18 years of age
* Symptomatic POP who desire vaginal or abdominal apical suspension
* English-speaking/reading
* Genital hiatus measurement < 6 cm, >2cm

Exclusion Criteria:

* Those who desire colpocleisis
* Those whose surgical planning includes levatorplasty
* Genital hiatus measurements greater than or equal to 6 cm, < 2 cm
* Inability to speak/understand English
* Those who specifically request a perineorrhaphy
* Pregnant patients

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2015-08 (Actual); Primary Completion 2017-05-01 (Actual); Study Completion 2017-05-01 (Actual)

PRIMARY OUTCOMES:
Body Image, by using the Body Image in Pelvic Organ Prolapse (BIPOP) questionnaire | 6 weeks post-operatively
  To determine if a patient's body image, by using the Body Image in Pelvic Organ Prolapse (BIPOP) questionnaire, is affected by concomitant performance of a perineorrhaphy at the time of pelvic organ prolapse surgery.

SECONDARY OUTCOMES:
Pelvic Organ Prolapse Quantification (POP-Q) Measurements | Pre-operatively, in the operating room, 1 week, 6 weeks, and 3 months post-operatively
  To determine if POP-Q measurements are affected by a perineorrhaphy, as measured immediately post-operatively, and at 1 week, 6 weeks and 3 months after surgery.
Pelvic Floor Muscle Strength as measured by the Peritron™ perineometer and digitally. | 6 weeks post-operatively
  To determine if the strength of pelvic floor muscles is improved after corrective pelvic organ prolapse surgery with a perineorrhaphy compared with those who did not have a perineorrhaphy, as measured by the Peritron™ perineometer and digitally.
Post-operative Pain by using a pain visual analog scale | 6 weeks post-operatively
  To assess if those having a perineorrhaphy have higher post-operative pain both in the short term and long term by using a pain visual analog scale both in the immediate and 6 week post-operative period.
Sexual Function, as measured by the validated questionnaire, PISQ-IR | 3 months post-operatively
  To describe if there are differences in sexual function after correction of pelvic organ prolapse with a perineorrhaphy compared to those that did not undergo a perineorrhaphy. The PISQ-IR is a validated questionnaire that measures sexual function in women with pelvic floor disorders in domains such as arousal, orgasm, partner-related issues, sexual quality, desire, and takes into account those who are not sexually active. The patients will fill out this questionnaire at a baseline visit and at post-operative visits.

CONTACTS AND LOCATIONS:
Overall Officials: Cara S Ninivaggio, MD, Principal Investigator — University of New Mexico
Locations (2):
- United States (2):
  - University of New Mexico, Albuquerque, New Mexico
  - Sandoval Regional Medical Center, Rio Rancho, New Mexico

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ninivaggio CS, Komesu YM, Jeppson PC, Cichowski SB, Qualls C, Qeadan F, Rogers RG, Dunivan GC. Perineorrhaphy Outcomes Related to Body Imagery: A Randomized Trial of Body Image Perception. Female Pelvic Med Reconstr Surg. 2021 May 1;27(5):281-288. doi: 10.1097/SPV.0000000000000841. PMID 32205557